CLINICAL TRIAL: NCT05067036
Title: The Effect of Physical Activity on Appetite and Food Intake in Older Adults
Brief Title: Physical Activity, Appetite and Food Intake in Older Adults (PHYSISAT)
Status: Completed | Type: Observational
Sponsor: University of Reading (Other)
Collaborators: Ministry of National Education, Turkey (Other Government)
Responsible Party: Principal Investigator, Miriam Clegg, Associate Professor, University of Reading
Other Study IDs: UREC 20/32
Record Dates: First submitted 2021-09-02; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2021-10

CONDITIONS: Older Adults; Physical Activity; Food Intake; Eating Behavior; Body Composition
Keywords: older adults; appetite; physical activity; food intake; body composition
MeSH Terms: conditions — Motor Activity; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the effect of physical activity on food intake and appetite in older adults (≥ 65 years) and to investigate the relationship between older adults' eating behaviours, body composition and physical activity.

DETAILED DESCRIPTION:
* To investigate the effect of physical activity on food intake and appetite in older adults (≥ 65 years).
* To examine the relationship between older adults' (≥ 65 years) eating behaviours, body composition and physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, living independently and self-reported;
* Aged ≥ 65 years;
* Having the ability to understand the study procedures.

Exclusion Criteria:

* Being obese (BMI > 30 kg/m2);
* Smoking more than 10 cigarettes a day;
* Having a disease such as cardiovascular disease and other chronic diseases (diabetes, thyroid disorders, cancer, heart, lung and kidney disease;
* Taking medications known to influence appetite, food intake or body weight in the past three months;
* Changing their diet and exercise in the last 3 months;
* Having unexpected weight loss in the last 3 months.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Participants aged older than 65 years.
Sampling Method: Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2020-12-09 (Actual); Primary Completion 2021-04-07 (Actual); Study Completion 2021-05-09 (Actual)

PRIMARY OUTCOMES:
Physical Activity Status | 7 days
  Physical Activity Status is assessed by using Accelerometers ((AX3) (3-Axis Logging Accelerometer)).
  Participants will wear the accelerometers 24-hour for 7 days. Their moderate and vigorous activity hours will be aggregated and based on this data, they will be divided into three groups as vigorous-moderate-low physical activity.
Ratings of Appetite | 1 day
  Appetite is assessed using a 100mm Visual Analogue Scales (VAS, scale 0-100).
Food Intake | 3 days (2 weekdays and 1 weekend day) while the participants are wearing the accelerometer.
  Food intake is assessed using a 24-hour weighted food diary.

SECONDARY OUTCOMES:
Height | Day 1
  Height is measured by using a tape measure.
Weight | Day 1
  Weight is assessed by using a body composition monitor (OMRON Viva).
BMI | Day 1
  BMI is assessed by using a body composition monitor (OMRON Viva).
% fat mass | Day 1
  % fat mass is assessed by using a body composition monitor (OMRON Viva).
% lean body mass | Day 1
  % lean body mass is assessed by using a body composition monitor (OMRON Viva).
Waist Circumference | Day 1
  Waist circumference is measured by using a tape measure.
Hip Circumference | Day 1
  Hip circumference is measured by using a tape measure.
Frailty | Day 1
  Frailty is assessed by using the 'Groingen Frailty Indicator Questionnaire'.
  The GFI is a validated, 15-item questionnaire with a score range from zero to fifteen that assesses the physical, cognitive, social, and psychological domains. A GFI score of four or greater is considered the cut-off point for frailty.
Nutritional Knowledge | Day 1
  Nutritional knowledge is assessed by using 'General Nutrition Knowledge Questionnaire'.
  This questionnaire consists of four independent sections, each assessing a different aspect of nutrition knowledge: Dietary recommendations; Food groups; Healthy Food choices and Diet, disease and weight management.
  Section 1 - Dietary Recommendations Each item carries one point for a correct answer. Maximum score = 18.
  Section 2 - Food groups Each item carries one point for a correct answer. Maximum score = 36
  Section 3- Healthy Food choices Each item carries one point for a correct answer. Maximum score = 13.
  Section 4 - Diet, disease and weight management Each item carries one point for a correct answer. Maximum score = 21.
Appetite Level based on 'Council on Nutrition Appetite Questionnaire' | Day 1
  Appetite level is assessed by using 'Council on Nutrition Appetite Questionnaire'.
  The score is calculated by adding up the points (values) that are assigned to the individual answers. The maximum number of points possible for a patient to obtain is 40, while the minimum is 8. The lower the score, the worse the patient's appetite.
  8-16: The patient is at risk for anorexia and needs nutrition counselling. 17-28: The patient needs frequent reassessment. >28: The patient is not at risk at this time.
Appetite Level based on 'The three-factor eating questionnaire' | Day 1
  Appetite level is assessed by using 'The three-factor eating questionnaire'.
  The TFEQ contains 51 items (questions) and measures three aspects of human eating behaviour: 'cognitive restraint of eating' (Factor I - 21 items); 'disinhibition' (Factor II - 16 items); 'hunger' (Factor III - 14 items). The minimum score for factors I-II-III is, therefore, 0-0-0, the possible maximum score 21-16-14.
Eating Behaviour | Day 1
  Eating behaviour is assessed by using the 'Dutch Eating Behaviour Questionnaire'
  The Dutch Eating Behavior Questionnaire is a 33-item self-report questionnaire to assess three distinct eating behaviours in adults: (1) emotional eating, (2) external eating, and (3) restrained eating. Items on the DEBQ range from 1 (never) to 5 (very often), with higher scores indicating greater endorsement of the eating behaviour.
Food Craving | Day 1
  The experience of food craving is assessed by using the 'Control of Eating Questionnaire'.
  The Control of Eating Questionnaire comprises 21-items that are designed to assess the severity and type of food cravings individual experiences over the previous 7 days. The overall score ranges from 0 to 200 and higher scores mean that they have higher severity of food cravings.
Physical Activity Level based on 'General Practice Physical Activity' questionnaire. | Day 1
  Physical activity level is assessed by using 'General Practice Physical Activity Questionnaire'.
  This questionnaire provides a simple, 4-level Physical Activity Index (PAI) of - Active, Moderately Active, Moderately Inactive, and Inactive.
  Inactive: Sedentary job and no physical exercise or cycling. Moderately inactive: Sedentary job and some but < 1 hour physical exercise and / or cycling per week OR Standing job and no physical exercise or cycling.
  Moderately active: Sedentary job and 1-2.9 hours physical exercise and / or cycling per week OR Standing job and some but < 1 hour physical exercise and / or cycling per week OR Physical job and no physical exercise or cycling.
  Active: Sedentary job and ≥ 3 hours physical exercise and / or cycling per week OR Standing job and 1-2.9 hours physical exercise and / or cycling per week OR Physical job and some but < 1 hour physical exercise and / or cycling per week OR Heavy manual job.
Physical Activity Level based on 'Physical Activity Scale for the Elderly (PASE)' questionnaire. | Day 1
  Physical activity level is assessed by using 'Physical Activity Scale for the Elderly (PASE)'.
  This questionnaire measures the level of self-reported physical activity in individuals aged 65 years or older and is considered of items regarding occupational, household, and leisure activities during the previous 7 day period. The total PASE score is computed by multiplying either the time spent in each activity (hours per week) or participation (i.e., yes/no) in an activity, by empirically derived item weights and then summing overall activities. The overall PASE score ranges from 0 to 400 or more.
Food shopping and cooking behaviors | Day 1
  Food shopping and cooking behaviors is assessed by using 'General Food Shopping and Cooking Questionnaire'.
  In this questionnaire, participant's food shopping and cooking behaviours will assess, no scale or score will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No personal identification data will be shared. The study is not under an obligation to share data, however, it is possible that some of the individual (unliked / non-identifiable) data will be useful in a meta-analysis and, hence sharing individual participant data (IPD) will be considered.

REFERENCES:
- [Background] Morley JE, Silver AJ. Anorexia in the elderly. Neurobiol Aging. 1988 Jan-Feb;9(1):9-16. doi: 10.1016/s0197-4580(88)80004-6. PMID 2898107
- [Background] Clegg ME, Godfrey A. The relationship between physical activity, appetite and energy intake in older adults: A systematic review. Appetite. 2018 Sep 1;128:145-151. doi: 10.1016/j.appet.2018.05.139. Epub 2018 Jun 7. PMID 29885385
- [Background] Clarkston WK, Pantano MM, Morley JE, Horowitz M, Littlefield JM, Burton FR. Evidence for the anorexia of aging: gastrointestinal transit and hunger in healthy elderly vs. young adults. Am J Physiol. 1997 Jan;272(1 Pt 2):R243-8. doi: 10.1152/ajpregu.1997.272.1.R243. PMID 9039015
- [Background] Margetts BM, Thompson RL, Elia M, Jackson AA. Prevalence of risk of undernutrition is associated with poor health status in older people in the UK. Eur J Clin Nutr. 2003 Jan;57(1):69-74. doi: 10.1038/sj.ejcn.1601499. PMID 12548299
- [Derived] Dericioglu D, Methven L, Clegg ME. Does physical activity level and total energy expenditure relate to food intake, appetite, and body composition in healthy older adults? A cross-sectional study. Eur J Nutr. 2025 Jan 24;64(2):71. doi: 10.1007/s00394-024-03571-z. PMID 39853478
- See also: NHS. 2018. Exercise as you get older — http://www.nhs.uk/live-well/exercise/exercise-as-you-get-older/
- See also: Age UK, Healthy eating — https://www.ageuk.org.uk/globalassets/age-ni/documents/information-guides/ageukig38_healthy_eating_inf.pdf